CLINICAL TRIAL: NCT05208918
Title: Effectiveness and Durability of Combined Application of Pulsed Radiofrequency and a Steroid to the Dorsal Root Ganglion for Postherpetic Neuralgia: a Randomized Controlled Trial
Brief Title: Combined Application of Pulsed RF and Steroids to the DRG for PHN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Collaborators: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mahmoud Mohammed Alseoudy, Lecturer of anesthesia, ICU & pain management; Faculty of Medicine, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZU-IRB#9199
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Postherpetic Neuralgia; Chronic Pain
MeSH Terms: conditions — Neuralgia, Postherpetic; Chronic Pain | interventions — Prolactin-Releasing Hormone; Steroids

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural steroid group (Active Comparator): Transforaminal steroid application to the dorsal root ganglion of the affected dermatome of herpes zoster related pain in affected patients
  Interventions: Procedure: Epidural steroid
- PRF plus steroids group (Active Comparator): Pulsed radiofrequency plus Depo-Medrol (steroid) application to the dorsal root ganglion of the affected dermatome of herpes zoster related pain in affected patients
  Interventions: Procedure: PRF plus steroids injection

INTERVENTIONS:
Procedure: Epidural steroid — Injection of Depo-Medrol of affected dermatomes
  Arms: Epidural steroid group
Procedure: PRF plus steroids injection — Pulsed radiofrequency with temperature 42 degrees for 6 minutes to be applied to the dorsal root ganglion plus injection of Depo-Medrol of affected dermatomes
  Arms: PRF plus steroids group

SUMMARY:
Recently, the use of pulsed radiofrequency has increased in many chronic pain conditions, including trigeminal neuralgia, chronic spinal pain, musculoskeletal pain, and it was recently used effectively for postherpetic neuralgia. Transforaminal epidural steroid injection has been proven in previous studies to provide effective analgesia for cases of herpes zoster-related pain. We hypothesize that the combined use of pulsed RF and steroid injection applied to the DRG may achieve better outcomes than the use of epidural steroid injection alone.

DETAILED DESCRIPTION:
Varicella-zoster virus reactivates in sensory ganglia as the dorsal root ganglion (DRG). The DRG contains many receptor channels and is an important region for pain signal transduction. Sustained abnormal electrical activity to the spinal cord via the DRG in acute herpes zoster can result in neuropathic conditions such as postherpetic neuralgia (PHN). Postherpetic neuralgia (PHN) is the final stage of varicella-zoster infection and is manifested as severe refractory neuropathic pain. Preventing the transition of herpes zoster-related pain to PHN is a very important therapeutic principle for patients at an early stage, especially for older patients. The exact discriminative time point for PHN has not yet been standardized. Various criteria have been used, from 30 days to 180 days after zoster onset. If pain persists for more than 180 days after zoster onset, the likelihood of pain reduction is very low and such a condition is considered "well established" PHN. Therefore, it is advisable to actively attempt various treatment modalities for pain control before the condition progresses to a recalcitrant state. Pulsed radiofrequency (PRF) is a variant of thermal radiofrequency that applies pulsed current to limit heat generation to less than 42˚C, creating a little risk of thermal or nerve injury. Recently, the use of PRF has increased in many chronic pain conditions, including trigeminal neuralgia, chronic spinal pain, musculoskeletal pain, and it was recently used effectively for postherpetic neuralgia. Transforaminal epidural steroid injection has been proven in previous studies to provide effective analgesia for cases of herpes zoster-related pain. We hypothesize that combined use of pulsed RF and steroid injection applied to the DRG may achieve a better outcome than use of epidural steroid injection alone.

ELIGIBILITY:
Inclusion Criteria:

* patients with ASA I&II status
* Thoracic zoster related pain
* less than three months duration from the appearance of shingles

Exclusion Criteria:

* coagulopathy
* local infection
* patient refusal
* Diabetes Melliteus

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale | Up to 6 months after the intervention
  Numerical rating scale (the 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable") to be recorded before intervention and at one week, 1 month , 2 months, and 3 months and 6 months after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud M Alseoudy, MD, Principal Investigator — mansoura university, faculty of medicine; khadega Elhossieny, MD, Study Director — Zagazig University
Locations (1):
- Zagazig university hospital, Zagazig, Ash-sharqia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang X, Li Y, Chen N, Zhou M, He L. Corticosteroids for preventing postherpetic neuralgia. Cochrane Database Syst Rev. 2023 Dec 5;12(12):CD005582. doi: 10.1002/14651858.CD005582.pub5. PMID 38050854